CLINICAL TRIAL: NCT06213389
Title: Comparison of EzVision® Videolaryngoscope and Gum Elastic Bougie-Assisted Machintosh Laryngoscopy in Patients Considering Difficult Intubation
Brief Title: Comparison of EzVision® Videolaryngoscope and Gum Elastic Bougie-Assisted Machintosh Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, MD, Principal Investigator, Nevsehir Public Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/1011
Record Dates: First submitted 2023-09-05; First posted 2024-01-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Intubation; Difficult or Failed; Airway Complication of Anesthesia
Keywords: Intubation; Difficult; Airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients to entubate with EzVision® videolaryngoscopy (Experimental): Patients will intubate with EzVision® videolaryngoscopy
  Interventions: Device: EzVision® videolaryngoscopy
- Patients to intubate with Macintosh blade (Other): Patients will intubate with Macintosh blade
  Interventions: Device: Macintosh Blade

INTERVENTIONS:
Device: EzVision® videolaryngoscopy — Patient will be intubated with EzVision® videolaryngoscopy
  Arms: Patients to entubate with EzVision® videolaryngoscopy
Device: Macintosh Blade — Patient will be intubated with Macintosh Blade
  Arms: Patients to intubate with Macintosh blade

SUMMARY:
The aim of this study is to compare the EzVision® videoryngoscope with conventional laryngoscopy using a Macintosh blade in patients with suspected difficult intubation. This study primarily aims to test the hypothesis that laryngoscopy image is better with EzVision® videoryngoscopy compared to direct laryngoscopy. The secondary hypothesis is also to test the view that, compared to direct laryngoscopy, EzVision® videolingoscopy will improve intubation success, reduce intubation attempts, shorten intubation time, facilitate intubation, and cause less additional complications such as bleeding or sore throat.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old;
2. American Association of Anesthesiologists (ASA) physical condition I-II-III;
3. Elective surgery requiring oral endotracheal intubation for general anesthesia;
4. Compliance with one of the difficult intubation estimation criteria (if more than one)
5. Expected extubation in the operating room

Exclusion Criteria:

1. Refusal to participate in research;
2. Age <18 and >65
3. ASA IV and above
4. Emergency cases
5. Body Mass Index (BMI) > 40 kg/m2.
6. Pregnancy
7. Cardiac surgery
8. Unexpectedly difficult intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Glottis viewing | Approximately 1 year
  Glottical viewing will be measured by Modified Cormack Lehane grading. In this scoring system, number 1 indicates the best appearance, while number 4 indicates the worst situation where the glottis is not visible. This measurement have no specific value, but it evaluates glottis opening as visually.
  1. Fill view of the glottis 2a. Partial view of the glottis 2b. Arytenoids or posterior part of the vocal cords only visible 3. Only epiglottis visible 4. Neither glottis nor epiglottis visible

SECONDARY OUTCOMES:
Intubation failure | Approximately 1 year
  Intubation failure: It is defined as intubation failure if one of the following occurs:
  * Failure to intubate despite three intubation attempts,
  * Situation that requires replacement of the intubation device,
  * Difficulty with intubation that will stop working at the discretion of the anesthesiologist
Attempted intubation | Approximately 1 year
  Attempted intubation: defined as inserting the endotracheal tube into the oral cavity to perform endotracheal intubation (Wang HE, Garza AG)
Intubation time | Approximately 1 year
  Intubation time: defined as the time between insertion of the laryngoscope into the oral cavity and the first appearance of end-tidal CO2.
  Ease of intubation: defined as the anesthetist's subjective assessment after finishing the intubation procedure as: (1) very easy; (2) easy; (3) medium; (4) difficult; and (5) impossible. (Ruetzler K) to.
Ease of intubation | Approximately 1 year
  Ease of intubation: defined as the anesthetist's subjective assessment after finishing the intubation procedure as: (1) very easy; (2) easy; (3) medium; (4) difficult; and (5) impossible. (Ruetzler K)

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

REFERENCES:
- [Result] Aziz MF, Dillman D, Fu R, Brambrink AM. Comparative effectiveness of the C-MAC video laryngoscope versus direct laryngoscopy in the setting of the predicted difficult airway. Anesthesiology. 2012 Mar;116(3):629-36. doi: 10.1097/ALN.0b013e318246ea34. PMID 22261795
- [Result] Butler PJ, Dhara SS. Prediction of difficult laryngoscopy: an assessment of the thyromental distance and Mallampati predictive tests. Anaesth Intensive Care. 1992 May;20(2):139-42. doi: 10.1177/0310057X9202000202. PMID 1595845
- [Result] Garza AG, Gratton MC, Coontz D, Noble E, Ma OJ. Effect of paramedic experience on orotracheal intubation success rates. J Emerg Med. 2003 Oct;25(3):251-6. doi: 10.1016/s0736-4679(03)00198-7. PMID 14585451
- [Result] Khan ZH, Kashfi A, Ebrahimkhani E. A comparison of the upper lip bite test (a simple new technique) with modified Mallampati classification in predicting difficulty in endotracheal intubation: a prospective blinded study. Anesth Analg. 2003 Feb;96(2):595-9, table of contents. doi: 10.1097/00000539-200302000-00053. PMID 12538218
- [Result] Lascarrou JB, Boisrame-Helms J, Bailly A, Le Thuaut A, Kamel T, Mercier E, Ricard JD, Lemiale V, Colin G, Mira JP, Meziani F, Messika J, Dequin PF, Boulain T, Azoulay E, Champigneulle B, Reignier J; Clinical Research in Intensive Care and Sepsis (CRICS) Group. Video Laryngoscopy vs Direct Laryngoscopy on Successful First-Pass Orotracheal Intubation Among ICU Patients: A Randomized Clinical Trial. JAMA. 2017 Feb 7;317(5):483-493. doi: 10.1001/jama.2016.20603. PMID 28118659
- [Result] Lewis SR, Butler AR, Parker J, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation. Cochrane Database Syst Rev. 2016 Nov 15;11(11):CD011136. doi: 10.1002/14651858.CD011136.pub2. PMID 27844477
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/22261795/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/1595845/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/14585451/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/12538218/